CLINICAL TRIAL: NCT04353830
Title: A Phase 1a, Open-label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Initial Efficacy of Recombinant Human Anti-T-cell Immunoreceptor With Ig and ITIM Domains (TIGIT) Monoclonal Antibody Injection (IBI939) in Subjects With Advanced Malignant Tumors
Brief Title: A Study Evaluating the Safety, Tolerability, and Initial Efficacy of Recombinant Human Anti-T-cell Immunoreceptor With Ig and ITIM Domains (TIGIT) Monoclonal Antibody Injection (IBI939) in Subjects With Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI939A101
Record Dates: First submitted 2020-04-17; First posted 2020-04-20 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ia Dose-Escalation Stage:IBI939 (Experimental): Participants will be treated with escalating doses of IBI939 to determine the MTD.
  Interventions: Drug: IBI939
- Phase Ia Dose-Escalation Stage:IBI939+ Sintilimab (Experimental): Participants will be treated with escalating doses of IBI939 in combination with a fixed dose of Sintilimab to determine the MTD.
  Interventions: Drug: IBI939+ Sintilimab
- Phase Ib Expansion Stage:IBI939+ Sintilimab (Experimental): Participants will be enrolled in the expansion stage to better characterize the safety, tolerability, PK variability, and preliminary efficacy of IBI939 in combination with Sintilimab in different cancer types.
  Interventions: Drug: IBI939+ Sintilimab

INTERVENTIONS:
Drug: IBI939 — Several dose levels will be evaluated for IBI939 administered as a single agent and in combination with Sintilimab. IBI939 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit. Those who discontinue treatment with single-agent IBI939 may receive combination treatment with Sintilimab or IBI939+ Sintilimab. Combination treatment may continue until disease progression or loss of clinical benefit.
  Arms: Phase Ia Dose-Escalation Stage:IBI939
Drug: IBI939+ Sintilimab — IBI939: Several dose levels will be evaluated for IBI939 in combination with Sintilimab. IBI939 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit.
  Sintilimab: Sintilimab will be given as 200 mg via IV infusion on Day 1 of each 21-day cycle in combination with IBI939. Combination treatment may continue until disease progression or loss of clinical benefit.
  Arms: Phase Ia Dose-Escalation Stage:IBI939+ Sintilimab
Drug: IBI939+ Sintilimab — IBI939: IBI939 in combination with Sintilimab will be given with RP2D. IBI939 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit.
  Sintilimab: Sintilimab will be given as 200 mg via IV infusion on Day 1 of each 21-day cycle in combination with IBI939. Combination treatment may continue until disease progression or loss of clinical benefit.
  Arms: Phase Ib Expansion Stage:IBI939+ Sintilimab

SUMMARY:
This is an open-label, dose escalation, Phase I study to evaluate the safety, tolerability, pharmacokinetics and efficacy of IBI939 in subjects with advanced malignancies

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF.
2. Adults 18 years of age or older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy at least 12 weeks.
5. Adequate organ and bone marrow function.

Eligibility Criteria：

1. Previous exposure to any anti-TIGIT antibody.
2. Participate in another interventional clinical study, except for the observational (non-interventional) clinical study or the survival follow-up phase of the interventional study.
3. Any investigational drugs received within 4 weeks prior to the first study treatment.
4. Receive the last dose of anti-tumor therapy within 4 weeks before the first dose of study therapy.
5. Immunosuppressive drugs were used within 4 weeks prior to the first administration of the study drug.
6. Medication requiring long-term systemic hormones or any other immunosuppression therapy.
7. Major surgical procedures (craniotomy, thoracotomy, or laparotomy) or unhealed wounds, ulcers, or fractures were performed within 4 weeks prior to the first dose of study therapy.
8. Primary central nervous system (CNS) malignancy, or untreated/active CNS metastases, or leptomeningeal disease.
9. History of autoimmune disease , present active autoimmune disease or inflammatory diseases
10. Positive human immunodeficiency virus (HIV) test.
11. Active hepatitis B or C, or tuberculosis.
12. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. Known history of hypersensitivity to any components of the IBI939 or Sintilimab.
14. Pregnant or nursing females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with AEs and SAEs | up to 2 years after enrollment
  To evaluate the safety and tolerability of IBI939 alone or in combination with Sintilimab [Adverse events (AEs), Serious Adverse Events (SAEs) ]
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | From Baseline to the end of Cycle 1
  To evaluate the safety and tolerability of IBI939 alone or in combination with Sintilimab.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | up to 2 years after enrollment
  The area under the curve (AUC) of serum concentration of the drug after the administration.
Pharmacokinetics: Cmax | up to 2 years after enrollment
  Maximum concentration (Cmax) of the drug after administration
Immunogenicity: Percentage of ADA positive subjects | up to 2 years after enrollment
  Immunogenicity: Number of Anti-Drug Antibodies (ADA) positive subjects will be counted and percentage of ADA positive subjects will be calculated to evaluate immunogenicity of IBI939.
Preliminary anti-tumor activity (Objective Response Rate) | up to 2 years after enrollment
  Objective Response Rate (ORR) is the percentage of Complete Response (CR) plus partial response (PR) assessed by RECIST v1.1 criteria for solid tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China